CLINICAL TRIAL: NCT02221765
Title: A Double-Blind, Randomised, Placebo-Controlled Dose Escalation Study to Assess the Safety, Tolerability and Efficacy of Single and Multiple Doses of PP 1420 in Healthy Subjects.
Brief Title: Safety, Tolerability and Efficacy Study of PP1420 in HV
Acronym: PP14201b1c
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Expected PK&no safety issues in 1B.1Cwon't proceed due to lack of 1Befficacy
Sponsor: Imperial College London (Other)
Collaborators: Wellcome Trust (Other); Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ICIM1420/14/01; 2014-001908-22 (EudraCT Number)
Record Dates: First submitted 2014-08-19; First posted 2014-08-20 (Estimated); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Obesity
Keywords: Obesity; Overnutrition; Nutrition Disorders; Overweight; Body Weight; Signs and Symptoms
MeSH Terms: conditions — Obesity; Overnutrition; Nutrition Disorders; Overweight; Body Weight; Signs and Symptoms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Visit 1 - sham visit: placebo 0.9% (w/v) saline single-dose, administered subcutaneously.
  Visit: 2 - placebo 0.9% (w/v) saline single-dose, administered subcutaneously.
  Visit 3 - single dose of PP 1420, administered subcutaneously. Dose levels: 8, 16, 32, 64 mg.
  Interventions: Drug: PP1420; Drug: Placebo
- Arm 2 (Experimental): Visit 1 - sham visit: placebo 0.9% (w/v) saline single-dose, administered subcutaneously.
  Visit: 2 - single dose of PP 1420, administered subcutaneously. Dose levels: 8, 16, 32, 64 mg.
  Visit 3 - placebo 0.9% (w/v) saline single-dose, administered subcutaneously.
  Interventions: Drug: PP1420; Drug: Placebo

INTERVENTIONS:
Drug: PP1420 — Single dose of PP 1420, administered subcutaneously. Dose levels: 8, 16, 32, 64 mg.
  Other Names: Pancreatic Polypeptide 1420
Drug: Placebo — 0.9% (w/v) saline single-dose, administered subcutaneously

SUMMARY:
Obesity is a growing pandemic which affects 1 in 4 adults in the UK, and shortens life by increasing cardiovascular disease, diabetes and cancer. Current treatments for obesity have either poor efficacy or significant side effects. Pancreatic polypeptide (PP) is a promising new drug target as it produces powerful appetite suppression which, following a 90-minute infusion continues to act for 24 h in man. We have developed a new long lasting high potency analogue of PP, PP1420. This is delivered as a once-a-day subcutaneous injection via a painless fine-gauge needle.

In a first-time-in-man Phase 1a trial, that PP 1420 proved safe, well tolerated, and had extended pharmacokinetics compared to PP itself.

We now plan to study the safety and PK of PP1420 up to 64mg. We will also assess:

1. Its efficacy in reducing food intake after a single dose in a Phase 1B study in healthy volunteers.
2. Its efficacy in reducing food intake and weight after multiple dosing in a Phase 1C study in healthy volunteers.

DETAILED DESCRIPTION:
More than 25% of people in the UK are obese. People with obesity have a shorter life expectancy, and have a higher risk of having heart attacks, strokes, high blood pressure, diabetes, and certain cancers.

At the moment, there is no treatment for obesity that is both effective and safe. Advising people to change their diet and to exercise more is frequently ineffective, and any loss in weight seen is usually temporary. There is only one medications licensed for the purpose of losing weight, but they are limited by side-effects. Finally, gastric bypass and similar surgeries are effective at reducing weight permanently, but can be risky and restricted only to very motivated people.

"Gut hormones" are natural chemicals made by the bowels when you eat. They work to reduce appetite and hunger when you eat, so that you will eat enough for your needs. We think that one of the reasons why gastric bypass surgery is so effective is because the surgery causes an increase in gut hormone secretion into the bloodstream, which suppresses appetite. One of these hormones is pancreatic polypeptide (PP), which is released into the bloodstream by cells in the pancreas after eating. When human PP is given to healthy volunteers as an injection, we see that they have a reduced appetite and food intake with no side-effects such as feeling sick or vomiting.

Human PP does not last long in the blood stream. In order to make it into a new, safe and effective drug for obesity, we have developed a new form of PP, which is very similar but not identical to human PP, that we expect will last longer in the blood. We call this PP 1420.

In testing, PP 1420 reduced food intake in animals, and was safe in them at much higher doses than those we plan to give in the current study.

PP1420 has previously been give to healthy volunteers in single doses up to 8mg without any serious problems. All doses were well tolerated.

This study will examine the safety and tolerability of PP 1420 when given at single doses of higher doses, up to 64 mg, and the safety, tolerability and efficacy of PP 1420 when given in multiple doses for up to 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male as determined by a responsible physician, based on a medical evaluation including history, physical examination, vital signs, laboratory tests and 12-lead ECG.
2. Between 18 and 50 years of age, inclusive, at the time of signing and dating the informed consent form.
3. Body weight 70 kg and body mass index (BMI) within the range 25 - 35 kg/m2 (inclusive).
4. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
5. Willing and able to comply with the protocol for the duration of the study.

Exclusion Criteria:

1. As a result of the medical interview, physical examination, or screening investigations, the Investigator considers the subject unsuitable for the study.
2. The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
3. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
4. A positive test for human immunodeficiency virus (HIV) antibody.
5. History of migraine.
6. History or evidence of abnormal eating behaviour, as observed through the Dutch Eating Behaviour (DEBQ) and SCOFF questionnaires.
7. History of excessive alcohol consumption within 6 months of the study defined as an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units. One unit is equivalent to 8 g of alcohol, a half-pint (approximately 240 mL) of beer or 1 measure (25 mL) of spirits or 1 glass (125 mL) of wine.
8. Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
9. Has QTc at screening >450 msec.
10. Systolic blood pressure outside the range 85 - 160 mmHg, diastolic blood pressure outside the range 45 - 100 mmHg, and/or heart rate outside the range 40 - 110 bpm.
11. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the dosing day in the current study: 90 days, five half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
12. Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
13. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 14 days or five half-lives (whichever is longer) prior to the dose of study medication, which, in the opinion of the Investigator, may interfere with the study procedures or compromise subject safety.
14. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator, contraindicates their participation.
15. Where participation in the study would result in donation of blood in excess of 500 mL within 3 months before or after the study.
16. Unwilling to abstain from:

    * Consumption of caffeine- or xanthine- containing products for 24 hours prior to dosing until the post-dose assessment at each treatment level.
    * Use of illicit drugs.
    * Alcohol for 48 hours prior to dosing until final post-dose assessment at each treatment level.
    * Smoking or otherwise consuming tobacco for 24 hours prior to dosing until the post-dose assessment at each treatment level.
17. Unwilling or unable to use a condom during sexual activity from first dose until the end of the study.
18. Vegans and subjects with milk or wheat intolerance or allergy as reported by the subject.
19. Unwillingness or inability to follow the procedures outlined in the protocol.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2014-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: | Within 7-10 days
  Safety and tolerability: adverse events (AEs); change from baseline in clinical chemistry, haematology and urine parameters; change from baseline outside the normal range for BP, heart rate, 12-lead electrocardiogram (ECG) parameters as specified below.

SECONDARY OUTCOMES:
Pharmacokinetic parameters | Within 7-10 days
  Pharmacokinetic parameters: AUC0-∞, AUC0-t, maximum observed plasma drug concentration (Cmax), time of maximum observed concentration (tmax), terminal elimination half-life (t½) and clearance.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bloom, Principal Investigator — Imperial College London
Locations (1):
- NIHR/ Wellcome Trust Imperial Clinical Research Facility, London, United Kingdom

REFERENCES:
- [Background] Batterham RL, Le Roux CW, Cohen MA, Park AJ, Ellis SM, Patterson M, Frost GS, Ghatei MA, Bloom SR. Pancreatic polypeptide reduces appetite and food intake in humans. J Clin Endocrinol Metab. 2003 Aug;88(8):3989-92. doi: 10.1210/jc.2003-030630. PMID 12915697
- [Background] Jesudason DR, Monteiro MP, McGowan BM, Neary NM, Park AJ, Philippou E, Small CJ, Frost GS, Ghatei MA, Bloom SR. Low-dose pancreatic polypeptide inhibits food intake in man. Br J Nutr. 2007 Mar;97(3):426-9. doi: 10.1017/S0007114507336799. PMID 17313701
- [Background] Tan TM, Field BC, Minnion JS, Cuenco-Shillito J, Chambers ES, Zac-Varghese S, Brindley CJ, Mt-Isa S, Fiorentino F, Ashby D, Ward I, Ghatei MA, Bloom SR. Pharmacokinetics, adverse effects and tolerability of a novel analogue of human pancreatic polypeptide, PP 1420. Br J Clin Pharmacol. 2012 Feb;73(2):232-9. doi: 10.1111/j.1365-2125.2011.04082.x. PMID 21834938